CLINICAL TRIAL: NCT01961453
Title: Targeting Wave Reflections to Improve Left Ventricular Hypertrophy, Fibrosis and Myocardial Function in Hypertension
Brief Title: Effect of Isosorbide Mononitrate on Hypertension to Improve Left Ventricular Hypertrophy, Fibrosis and Myocardial Function
Acronym: ISMN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01442
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
Keywords: Hypertension; Isosorbide Mononitrate; Myocardial fibrosis
MeSH Terms: conditions — Hypertension | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isosorbide Mononitrate, sustained release (Active Comparator): One tablet containing 60 mg (Titration Stage 1) OR 120 mg (Titration Stage 2) of sustained-release ISMN administered at 8 AM.
  Interventions: Drug: Isosorbide Mononitrate, sustained release
- Placebo capsule (Placebo Comparator): One capsule of placebo administered once daily at 8 AM
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Isosorbide Mononitrate, sustained release — 60 mg if Titration Stage 1 OR 120 mg if Titration Stage 2
  Arms: Isosorbide Mononitrate, sustained release
Drug: Placebo capsule — One capsule of placebo administered once daily at 8 am.
  Arms: Placebo capsule

SUMMARY:
The purpose of this research study is to test whether treatment with isosorbide mononitrate will improve left ventricular hypertrophy ("thickening") which puts people at risk for developing heart failure. Once it develops, heart failure is a very serious condition and thus it is important to find ways to prevent it from happening. The investigators have reasons to believe that dilating the blood vessels with this specific medication will improve the thickening of the heart, which increases the risk of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure >140 mmHg, diastolic blood pressure > 90 mmHg.
* An elevated left ventricular mass index (defined as >60 g/m1.7 in women and 80 g/m1.7 in men) OR LV posterior wall thickness >1.4 cm documented in a clinically indicated echocardiographic examination or magnetic resonance imaging scan within the previous 12 months.
* Stable medical therapy as defined by: (1)No addition or removal of ACE inhibitors, angiotensin receptor blockers, beta-blockers, or calcium channel blockers for 30 days. (2)No change in dosage of ACE, angiotensin-receptor blocker, beta-blockers or calcium-channel blockers s of more than 100% for 30 days.
* Current therapy with an ACE inhibitor, hydralazine or a statin, all of which have been shown to reduce nitrate tolerance.

Exclusion Criteria:

* Rhythm other than sinus rhythm (i.e., atrial fibrillation).
* Non-cardiac condition limiting life expectancy to less than one year, per physician judgment.
* Current or anticipated future need for nitrate therapy.
* Valve disease (> mild aortic or mitral stenosis; > moderate aortic or mitral regurgitation).
* Hypertrophic cardiomyopathy.
* Known infiltrative or inflammatory myocardial disease (amyloid, sarcoid).
* Pericardial disease.
* Primary pulmonary arteriopathy.
* Have experienced a myocardial infarction or unstable angina, or have undergone percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) within 60 days prior to consent, or requires either PTCA or CABG at the time of consent.
* Resting heart rate (HR) > 100 bpm.
* A reduced LV ejection fraction (EF<50%).
* Known severe liver disease (AST > 3x normal, alkaline phosphatase or bilirubin > 2x normal).
* Patients with a clinically indicated stress test demonstrating significant ischemia within a year of enrollment which was not followed by percutaneous or surgical revascularization.
* Allergy to isosorbide mononitrate.
* Current therapy with phosphodiesterase inhibitors, such as sildenafil, vardenafil or tadalafil, since the combination of nitrates and phosphodiesterase inhibitors can result in severe hypotension.
* Therapy with rosiglitazone, since this combination is not recommended based on epidemiologic data suggesting that it may increase the risk of myocardial ischemia.
* Current pregnancy or a positive urine pregnancy test. Women who become pregnant during the study will be discontinued from the trial.
* Contraindications to a cardiac MRI: (i) Central nervous system aneurysm clips; (ii) Implanted neural stimulators; (iii) Implanted cardiac pacemaker or defibrillator; (iv) Cochlear implant; (v) Ocular foreign body (e.g. metal shavings); (vi) Other implanted medical devices: (e.g. drug infusion ports); (vii) Insulin pump; (viii) Metal shrapnel or bullet; (ix) Claustrophobia; (x) Extreme obesity rendering the patient unable to fit into narrow-bore scanners; (xi) Unwillingness of the patient to undergo a cardiac MRI. All patients with metallic implants will be individually evaluated prior to MRI.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass | 24 weeks

SECONDARY OUTCOMES:
Change in extracellular volume fraction | 24 weeks
Change in peak myocardial systolic longitudinal strain measured by MRI | 24 weeks
Change in peak early diastolic intraventricular pressure gradient measured by MRI | 24 weeks
Change in late systolic hypertension derived from pulse wave analysis | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Chirinos, MD, PhD, Principal Investigator — Philadelphia VA Medical Center & University of Pennsylvania
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bradley JG, Davis KA. Orthostatic hypotension. Am Fam Physician. 2003 Dec 15;68(12):2393-8. PMID 14705758
- [Background] Li H, Wang SX. Improvement of hypertension and LVH in maintenance hemodialysis patients treated with sustained-release isosorbide mononitrate. J Nephrol. 2011 Mar-Apr;24(2):236-45. doi: 10.5301/jn.2011.6252. PMID 21240870